CLINICAL TRIAL: NCT05236192
Title: Navy and Marine Corps New Parent Support Program Evaluation
Brief Title: New Parent Support Program Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ryan Chesnut, Assistant Research Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00019356
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-01

CONDITIONS: Child Maltreatment

STUDY DESIGN:
Intervention Model Description: A cluster randomized control trial effectiveness-implementation hybrid type 2 design will be used. Navy and Marine Corps installations participating in this study will be randomly assigned to one of two conditions: TRHV and SAU. Families receiving NPSP home visiting services will be administered TRHV or SAU depending upon the assignment of their installation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Take Root Home Visitation (TRHV) (Experimental): TRHV is an evidence-informed, manualized home-visiting curriculum.
  Interventions: Behavioral: Take Root Home Visitation (TRHV)
- Services as Usual (SAU) (Active Comparator): SAU involves the current standard of care implemented at the participating Navy and Marine Corps installations.
  Interventions: Behavioral: Services as Usual (SAU)

INTERVENTIONS:
Behavioral: Take Root Home Visitation (TRHV) — TRHV is a home-visiting, standardized program that home visitors can use to structure their time spent with families during home visits.
  Arms: Take Root Home Visitation (TRHV)
Behavioral: Services as Usual (SAU) — SAU includes an installation's current NPSP home visiting practice, which may vary across the installations participating in this study.
  Arms: Services as Usual (SAU)

SUMMARY:
The purpose of this study is to perform a program evaluation of the Navy and Marine Corps' New Parent Support Program (NPSP) home-visiting option. Both the Navy and Marine Corps have decided to pilot the Take Root Home Visitation (TRHV) curriculum, which is an evidence-informed, standardized program, with clients receiving NPSP home visits. This study is designed to examine the implementation and program effectiveness of TRHV compared to services as usual (SAU). Program outcomes include child development, parenting behaviors, child maltreatment risk and protective factors, and child maltreatment incidents. Implementation outcomes include clinicians' and clients' satisfaction with the program, clinicians' fidelity to the program delivery model, and clients' engagement with the program.

DETAILED DESCRIPTION:
The Navy and Marine Corps' NPSP home visiting option assists families who are at risk for child abuse and neglect by providing those families with home visitation by a trained professional (e.g., licensed clinical social worker, nurse). The ultimate goal of NPSP home visiting is to promote strong parenting practices and healthy families by providing parents with skills to foster child development and well-being. Families, expecting a child and with children up to age three, participating in the NPSP home visiting services at select military installations will be recruited for a cluster randomized controlled effectiveness-implementation hybrid Type 2 design program evaluation, which simultaneously tests the implementation and client related outcomes of a program (Curran et al., 2012).

Rigorous program evaluations of Navy and Marine Corps NPSP home visiting services are lacking. In fact, only one published study evaluating Navy NPSP could be located (Kelley et al., 2006). While the results of Kelley et al.'s (2006) study were generally positive, it was a single-group retrospective design that did not assess implementation outcomes or program outcomes related to child maltreatment. Thus, that study's ability to inform NPSP home visiting services is limited. Further, findings from past analyses of Army NPSP offered no evidence that NPSP services directly prevent child abuse and neglect (Kaye, Faber, Schiavone, & Perkins, 2016). Among the general U.S. population, research findings are mixed with regard to the effectiveness of home visiting programs for preventing child maltreatment (Howard & Brooks-Gunn, 2009; Kaminski, Valle, Filene, & Boyle, 2008). However, the available evidence does indicate that these programs can positively alter parenting practices.

Without a rigorous, experimental evaluation, it is difficult to assess whether the Navy's and Marine Corps' NPSP service as usual (SAU) is having the intended impacts on participating families. Further, the both Services are interested in exploring the utility of delivering the Take Root Home Visitation (TRHV) program. TRHV is a newly developed, evidence-informed, secondary, home-visiting prevention program developed by researchers at the Clearinghouse for Military Family Readiness at Penn State in collaboration with the Office of the Deputy Assistant Secretary of Defense for Military Community and Family Policy. TRHV has not been evaluated within the context of the Navy or Marine Corps. TRHV has been implemented with the Army as part of the Clearinghouse's three-phase evaluation of Army NPSP. Though the final report is still forthcoming, a preliminary report on program implementation showed that home visitors found TRHV to be acceptable and were able to implement the program with fidelity (Kaye et al., 2021). Moreover, parents receiving TRHV reported high levels of satisfaction with the program and stayed in NPSP services longer than parents receiving SAU (Kaye et al., 2021).

The extent to which the Army TRHV implementation findings generalize to the Navy and Marine Corps is unclear. Additionally, it is unclear to what extent TRHV will impact program outcomes, especially when compared to SAU. This study is designed to help bring clarity to these issues.

ELIGIBILITY:
Inclusion Criteria (NPSP Participants):

* 18+ years old
* Stationed at one of the participating military installations
* Active duty, retired, National Guard or Reserves service member or spouse/partner
* Pregnant or have a child 0-3-years-old
* Eligible to receive NPSP home-visiting services
* Speak and understand English proficiently

Inclusion Criteria (NPSP Home Visitors):

* 18+ years old
* Working at one of the participating military installations as a NPSP home visitor
* Speak and understand English proficiently

Inclusion Criteria (NPSP Participants' Children):

* Children of active duty, retired, National Guard or Reserves service member or spouse/partner receiving NPSP home-visiting services
* 0-3-years-old

Exclusion Criteria (NPSP Participants):

* Younger than 18 years of age
* Not stationed at one of the participating military installations
* Not an active duty, retired, National Guard or Reserves service member or spouse/partner
* Not currently pregnant or the parent of a child 0-3-years-old
* Not eligible for NPSP home-visiting services
* Does not speak or understand English proficiently

Exclusion Criteria (NPSP Home Visitors):

* Younger than 18 years of age
* Not employed at one of the participating military installations as a NPSP home visitor
* Does not speak or understand English proficiently

Exclusion Criteria (NPSP Participants' Children):

* Not the child of an active duty, retired, National Guard or Reserves service member or spouse/partner receiving NPSP home-visiting services
* Older than 3 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Change in Brief Child Abuse Potential Inventory (BCAP) | Baseline, 3-4 months post-baseline, 6-7 months post-baseline, and NPSP service or study completion (whichever occurs first - study completion is approximately 12 months post-baseline)
  The BCAP is the short form of the Child Abuse Potential Inventory (CAPI), which assesses potential risk for child abuse. Scores range from 0-24 with higher scores indicating greater risk.
Child Maltreatment Incident Report | Study completion, which is approximately 12 months post-baseline
  Administrative data will be collected to determine if a child maltreatment incident has occurred.
Change in Ages & Stages Questionnaire, Third Edition (ASQ-3) | Baseline, 3-4 months post-baseline, 6-7 months post-baseline, and NPSP service or study completion (whichever occurs first - study completion is approximately 12 months post-baseline)
  ASQ-3 is a standardized measure of child development across five domains: communication, gross motor, fine motor, problem-solving, and personal-social. Questionnaires are based on child age (and prematurity status). Scores range from 0-60 within each domain with higher scores reflecting typical development. Raw scores within each domain are classified into typical development, monitoring, and referral categories based upon established cut-off criteria.
Change in Parenting Skills Assessment 10th Edition (PSA-10) | Baseline, 6-7 months post-baseline, and NPSP service or study completion completion (whichever occurs first - study completion is approximately 12 months post-baseline)
  PSA-10 is an observational tool designed to measure parenting skills across five domains: communication with child, child management and supervision, parent/child activities, nurturing, and enriched environment. Domain scores range from 5 to 20 with higher scores indicating greater competence in that skill area.
Change in Family Needs Screener (FNS) | Baseline, 6-7 months post-baseline, and NPSP service or study completion completion (whichever occurs first - study completion is approximately 12 months post-baseline)
  FNS is a family violence risk screener that assess 10 factors: demographics, stress, relationship discord, support, substance abuse, violence approval, family of origin violence and neglect, self-esteem, depression, and prior family violence. Scores for item scale item are dichotomized and summed such that total scores range from 0 to 53 with a score of 9 or higher being classified as high needs.
Change in Protective Factors Survey (PFS) | Baseline, 6-7 months post-baseline, and NPSP service or study completion completion (whichever occurs first - study completion is approximately 12 months post-baseline)
  PFS assesses the presence of factors known to buffer against child maltreatment, such as family functioning, emotional support, concrete support, and nurturing and attachment. Subscale scores range from 1 to 7 with higher scores reflecting greater protection.
Change in Parental Stress Scale (PSS) | Baseline, 3-4 months post-baseline, 6-7 months post-baseline, and NPSP service or study completion (whichever occurs first - study completion is approximately 12 months post-baseline)
  PSS assesses four aspects of parenting stress: parental rewards, parental stressors, lack of control, and parental satisfaction. Subscale scores can be computed, but most often, a total score, ranging from 18 (low stress) to 90 (high stress), is calculated.
Change in Center for Epidemiological Studies Depression Scale (CESD-10) | Baseline, 6-7 months post-baseline, and NPSP service or study completion completion (whichever occurs first - study completion is approximately 12 months post-baseline)
  CESD-10 is a brief measure that assesses depressive symptoms over the prior week. Scores range from 0 to 30, with higher scores indicating greater depression.
Client Satisfaction Questionnaire (CSQ-8) | 6-7 months post-baseline and NPSP service or study completion completion (whichever occurs first - study completion is approximately 12 months post-baseline)
  CSQ-8 measures clients' satisfaction with the services they have received. Scores range from 8 to 32 with higher scores reflecting greater satisfaction.
Client Engagement Survey (CES) | 3-4 months post-baseline, 6-7 months post-baseline, and NPSP service or study completion (whichever occurs first - study completion is approximately 12 months post-baseline)
  CES is a measure of clients' engagement with the services they are receiving. Four domains of engagement are assessed: receptivity (score range: 4 to 20), buy-in (score range: 9 to 40), working relationship (score range: 4 to 20), and mistrust (score range: 3 to 15). The total engagement score ranges from 20 to 95 with higher scores reflecting greater engagement.
Evidence-Based Practice Attitude Scale (EBPAS) | Baseline
  EBPAS assesses providers' attitudes regarding the adoption of new treatments, interventions, and practices. Four domains are measured: requirements, appeal, openness, and divergence. Subscale scores and the total score are calculated by averaging the appropriate items, so scores range from 0 to 4 with higher scores indicating more of the construct of interest.
Treatment Fidelity | Baseline, 3-4 months post-baseline, 6-7 months post-baseline, and NPSP service or study completion (whichever occurs first - study completion is approximately 12 months post-baseline)
  Brief checklists will be used to assess NPSP home visitors' adherence to the program model.

SECONDARY OUTCOMES:
Program Reach | Study completion, which is approximately 12 months post-baseline
  Family Advocacy Program (FAP) managers will be asked to provide the percentage of eligible families who received TRHV and SAU.
Program Penetration | Study completion, which is approximately 12 months post-baseline
  FAP managers will be asked to provide the percentage of eligible home visitors who delivered TRHV and SAU.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan P Chesnut, PhD, Principal Investigator — The Pennsylvania State University; Daniel F Perkins, PhD, Principal Investigator — The Pennsylvania State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Kelley, M. L., Schwerin, M. J., Farrar, K. L., & Lane, M. E. (2006). A participant evaluation of the U.S. Navy parent support program. Journal of Family Violence, 21, 301-310. https://doi.org/10.1007/s10896-006-9031-5
- [Background] Kaye, M. P., Faber, A., Schiavone, W., & Perkins, D. F. (2016). New Parent Support Program Engagement Phase II Final Report. University Park, PA: Clearinghouse for Military Family Readiness at Penn State.
- [Background] Kaye, M. P., Ferrara, A. M., Abram-Erby, G., Kotch, R., Gernon, S., & Perkins, D. F. (2021, April). Take Root Home Visitation implementation: Army New Parent Support Program (NPSP) EIII. University Park, PA: Clearinghouse for Military Family Readiness at Penn State.
- [Background] Kaminski JW, Valle LA, Filene JH, Boyle CL. A meta-analytic review of components associated with parent training program effectiveness. J Abnorm Child Psychol. 2008 May;36(4):567-89. doi: 10.1007/s10802-007-9201-9. Epub 2008 Jan 19. PMID 18205039
- [Background] Howard KS, Brooks-Gunn J. The role of home-visiting programs in preventing child abuse and neglect. Future Child. 2009 Fall;19(2):119-46. doi: 10.1353/foc.0.0032. PMID 19719025